CLINICAL TRIAL: NCT00217438
Title: A Multi-Center Phase III Study of Autologous Transplantation for Patients With Multiple Myeloma Comparing Melphalan 280 mg/m2 + Amifostine With Melphalan 200 mg/m2 + Amifostine
Brief Title: Melphalan and Amifostine Followed By One or Two Autologous or Syngeneic Stem Cell Transplants and Maintenance Therapy in Treating Patients With Stage II-III Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004.00; NCI-2009-01543 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Refractory Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Amifostine; Peripheral Blood Stem Cell Transplantation; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (high dose melphalan, amifostine trihydrate, transplant) (Experimental): INDUCTION THERAPY:
  Patients receive amifostine IV over 3-5 minutes on days -3 and -2 followed by high-dose melphalan IV over 15-30 minutes on day 2.
  AUTOLOGOUS OR SYNGENEIC PBSCT: At least 20 hours after completion of melphalan, patients undergo autologous or syngeneic PBSCT on day 0.
  Patients undergo restaging of the disease between days 80-90. Patients with progressive disease are removed from the study. Patients who achieve a CR or near-CR can proceed to optional maintenance therapy. Patients who do not achieve a CR or near-CR may undergo additional induction therapy as in arm I followed by a second autologous or syngeneic PBSCT.
  Patients again undergo restaging of the disease 80-90 days later. Patients with progressive disease are removed from the study. Patients without progressive disease can proceed to maintenance therapy.
  Interventions: Drug: melphalan; Drug: amifostine trihydrate; Procedure: peripheral blood stem cell transplantation; Genetic: fluorescence in situ hybridization; Procedure: bone marrow ablation with stem cell support
- Arm II (low dose melphalan, amifostine trihydrate, transplant) (Active Comparator): INDUCTION THERAPY:
  Patients receive amifostine as in arm I and melphalan as in arm I at a lower dose.
  AUTOLOGOUS OR SYNGENEIC PBSCT: At least 20 hours after completion of melphalan, patients undergo autologous or syngeneic PBSCT on day 0.
  Patients undergo restaging of the disease between days 80-90. Patients with progressive disease are removed from the study. Patients who achieve a CR or near-CR can proceed to optional maintenance therapy. Patients who do not achieve a CR or near-CR may undergo additional induction therapy as in arm I followed by a second autologous or syngeneic PBSCT.
  Patients again undergo restaging of the disease 80-90 days later. Patients with progressive disease are removed from the study. Patients without progressive disease can proceed to maintenance therapy.
  Interventions: Drug: melphalan; Drug: amifostine trihydrate; Procedure: peripheral blood stem cell transplantation; Genetic: fluorescence in situ hybridization; Procedure: bone marrow ablation with stem cell support

INTERVENTIONS:
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Drug: amifostine trihydrate — Given IV
  Other Names: ethiofos; Ethyol; gammaphos; WR-2721
Procedure: peripheral blood stem cell transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Genetic: fluorescence in situ hybridization — Correlative study
  Other Names: fluorescence in situ hybridization (FISH)
Procedure: bone marrow ablation with stem cell support — Undergo transplant

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy. Giving chemotherapy with a peripheral stem cell transplant once or twice, using stem cells from the patient or an identical brother or sister, may allow more chemotherapy to be given so more cancer cells are killed. Giving maintenance therapy after a stem cell transplant may kill any cancer cells that remain. It is not yet known which dose of melphalan is more effective in treating multiple myeloma (MM).

PURPOSE: This randomized phase III trial is studying two different doses of melphalan to compare how well they work when given together with amifostine followed by one or two autologous or syngeneic stem cell transplants and maintenance therapy in treating patients with stage II-III MM

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the complete response (CR) and near CR rate in patients undergoing autologous stem cell transplant (ASCT) using melphalan 280 mg/m^2 or melphalan 200 mg/m^2.

SECONDARY OBJECTIVES:

I. Compare toxicities between patients receiving amifostine and melphalan 280 mg/m^2 or melphalan 200 mg/m^2.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

INDUCTION THERAPY:

ARM I (HIGH DOSE MELPHALAN AND AMIFOSTINE): Patients receive amifostine intravenously (IV) over 3-5 minutes on days -3 and -2 followed by high-dose melphalan IV over 15-30 minutes on day 2.

ARM II (LOW DOSE MELPHALAN AND AMIFOSTINE): Patients receive amifostine as in arm I and melphalan as in arm I at a lower dose.

AUTOLOGOUS OR SYNGENEIC PERIPHERAL BLOOD STEM CELL TRANSPLANTATION (PBSCT): At least 20 hours after completion of melphalan, patients undergo autologous or syngeneic PBSCT on day 0.

Patients undergo restaging of the disease between days 80-90. Patients with progressive disease are removed from the study. Patients who achieve a CR or near-CR can proceed to optional maintenance therapy. Patients who do not achieve a CR or near-CR may undergo additional induction therapy as in arm I followed by a second autologous or syngeneic PBSCT.

Patients again undergo restaging of the disease 80-90 days later. Patients with progressive disease are removed from the study. Patients without progressive disease can proceed to maintenance therapy.

After completion of study treatment, patients are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have MM undergoing autologous or syngeneic hematopoietic transplantation
* Patients must meet Salmon and Durie criteria for initial diagnosis of MM
* Transplant will be offered to patients with stage II or III MM
* Measurable disease, defined as serum monoclonal protein >= 0.2 g/dl or Bence Jones protein >= 200 mg/24 h
* Karnofsky >= 70 or Eastern Cooperative Oncology Group (ECOG) 0-2
* Life expectancy is not severely limited by concomitant illness
* Left ventricular ejection fraction >= 50%
* No uncontrolled arrhythmias or symptomatic cardiac disease
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and diffusion capacity of carbon monoxide (DLCO) >= 50%
* No symptomatic pulmonary disease
* Human immunodeficiency virus (HIV) negative
* Bilirubin < 2 mg/dl
* Serum glutamic pyruvate transaminase (SGPT) < 2.5 x normal
* Creatinine clearance >= 60 cc/min, estimated or measured
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating females
* Uncontrolled infection
* Planned tandem autologous/reduced intensity allograft
* Insufficient PBSC for an autologous transplant (< 3.0 x 10^6 CD34+ cells/kg total)
* Prior autologous transplant
* Non-secretory myeloma and patients who are in a complete response or near complete response after conventional therapy
* Patients unwilling to practice adequate forms of contraception if clinically indicated
* Male patients on study need to be consulted to use latex condoms, even if they have had a vasectomy, every time they have sex with a woman who is able to have children
* Patients with history of seizures
* Patients receiving antihypertensive therapy that cannot be stopped for 24 hours preceding amifostine treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-07; Primary Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bensinger, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Rochester, Rochester, New York
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial opened for enrollment September 2005 and completed enrollment in June 2012. Patients were enrolled at 4 centers: University of Washington, Seattle, WA; Veteran's Administration Puget Sound Healthcare Administration, Seattle, WA; Cedars Sinai Medical Center, Los Angeles, CA; and James Wilmot Cancer Center in Rochester, NY.
Period: Overall Study
Arm/Group | Arm I (High Dose Melphalan, Amifostine Trihydrate, Transplant) | Arm II (Low Dose Melphalan, Amifostine Trihydrate, Transplant)
Started | 66 | 64
Completed | 66 | 63 (One patient did not complete Day 80-120 evaluation tests after returning to referring physician.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (High Dose Melphalan, Amifostine Trihydrate, Transplant) | Arm II (Low Dose Melphalan, Amifostine Trihydrate, Transplant) | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 55 | 112
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 43 | 41 | 84
Region of Enrollment [Number; unit: participants]
  United States | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: CR and Near CR Rates
Description: Per modified European Group for Blood and Marrow Transplant (EBMT) response criteria for definition of response in patients with multiple myeloma treated by high-dose therapy and stem cell transplantation: Complete Response (CR): Complete disappearance of all clinically measurable disease, complete response requires negative tests for monoclonal proteins in serum and urine by immunofixation, no monoclonal plasma cells in marrow specimen by flow cytometry and no evidence of progressive bone disease by skeletal survey. "Near" Complete Response (nCR): Less than 0.1 gram/dL monoclonal protein detectable in serum by standard protein electrophoresis and less than 50 mg monoclonal protein detectable in urine on 24 hour collection. Less than 5% monoclonal plasma cells detectable in bone marrow by immunohistochemistry. No evidence of progressive bone disease by skeletal survey.
Time Frame: Up to 120 days after transplant
Population: Per protocol, patients who completed the day 80-120 evaluation assessments.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (High Dose Melphalan, Amifostine Trihydrate, Transplant) | Arm II (Low Dose Melphalan, Amifostine Trihydrate, Transplant)
Number analyzed (Participants) | 66 | 63
percentage of participants | 39 | 22

2. Secondary Outcome: Relative Toxicities Between Melphalan 280 mg/m^2 or Melphalan 200 mg/m^2
Description: Number of Grade 3-4 adverse events observed in each group from enrollment through the Day 80-120 evaluation. Grade 3-4 events are defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: Up to day 56 after transplant
Population: Patients who were treated per protocol.
Measure: Number; unit: Grade 3-4 adverse events
Arm/Group | Arm I (High Dose Melphalan, Amifostine Trihydrate, Transplant) | Arm II (Low Dose Melphalan, Amifostine Trihydrate, Transplant)
Number analyzed (Participants) | 66 | 64
Grade 3-4 adverse events | 20 | 10

ADVERSE EVENTS:
Arm/Group | Arm I (High Dose Melphalan, Amifostine Trihydrate, Transplant) | Arm II (Low Dose Melphalan, Amifostine Trihydrate, Transplant)
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/64
Other Adverse Events (participants affected / at risk) | 14/66 | 7/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (High Dose Melphalan, Amifostine Trihydrate, Transplant) (N=66) | Arm II (Low Dose Melphalan, Amifostine Trihydrate, Transplant) (N=64)
Mucositis-Grade 3 or higher (Gastrointestinal disorders) | 7 (7) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 3 (3) — Mucositis recorded separately.
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenic fever (Nervous system disorders) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 7 (7) | 2 (2) — Mucositis recorded separately
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Graft versus host disease of the gut (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication. In the event the sponsor decides a patent application should be filed, the embargo may extend up to an additional 60 days or until a patent application is filed.